CLINICAL TRIAL: NCT05493657
Title: Aspirin Versus Clopidogrel for Leaflet Thrombosis Prevention in Patients Undergoing Transcatheter Aortic Valve Replacement: ACLO-TAVR Trial
Brief Title: Aspirin vs Clopidogrel After TAVR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2022-0744
Record Dates: First submitted 2022-08-08; First posted 2022-08-09 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Severe Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin group (Active Comparator): Patients receive the aspirin (100 mg/day) single antiplatelet therapy after 4 weeks of dual antiplatelet therapy of aspirin (100 mg/day) and clopidogrel (75 mg/day) after TAVR.
  Interventions: Drug: Aspirin single antiplatelet therapy
- Clopidogrel group (Experimental): Patients receive the clopidogrel (75 mg/day) single antiplatelet therapy after 4 weeks of dual antiplatelet therapy of aspirin (100 mg/day) and clopidogrel (75 mg/day) after TAVR.
  Interventions: Drug: Clopidogrel single antiplatelet therapy

INTERVENTIONS:
Drug: Aspirin single antiplatelet therapy — Patients receive the aspirin (100 mg/day) single antiplatelet therapy after 4 weeks of dual antiplatelet therapy of aspirin (100 mg/day) and clopidogrel (75 mg/day) after TAVR.
  Arms: Aspirin group
Drug: Clopidogrel single antiplatelet therapy — Patients receive the clopidogrel (75 mg/day) single antiplatelet therapy after 4 weeks of dual antiplatelet therapy of aspirin (100 mg/day) and clopidogrel (75 mg/day) after TAVR.
  Arms: Clopidogrel group

SUMMARY:
Currently, the optimal antithrombotic therapy after transcatheter aortic valve replacement (TAVR) remains still unknown., The purpose of the study is to compare aspirin versus clopidogrel monoantiplatelet therapy for preventive effect on leaflet thrombosis in patients undergoing TAVR for severe aortic stenosis. This study is designed as a prospective, multicenter, open label, randomized controlled study. Eligible patients will be randomized to aspirin or clopidogrel monotherapy after TAVR. Patients will have dual antiplatelet therapy of aspirin 100 mg and clopidogrel 75 mg for 4 weeks after TAVR and then subsequent monoantiplatelet therapy of either aspirin 100 mg or clopidogrel 75 mg according to the randomization. Leaflet thrombosis will be assessed with cardiac computed tomography (CT) and transthoracic echocardiography at 3 months after TAVR. Patients will be clinically followed for 6 months. The primary endpoint is the Incidence of leaflet thrombosis on cardiac CT at 3 months.

DETAILED DESCRIPTION:
1. Prospective, multicenter, open label, randomized controlled study
2. Eligible patients will be randomized to aspirin or clopidogrel monotherapy after TAVR
3. All patients will have dual antiplatelet therapy of aspirin 100 mg and clopidogrel 75 mg for 4 weeks after TAVR and then subsequent monoantiplatelet therapy of either aspirin 100 mg or clopidogrel 75 mg.
4. Leaflet thrombosis will be assessed with cardiac computed tomography (CT) and transthoracic echocardiography at 3 months after TAVR
5. Clinical follow-up up to 6 months

ELIGIBILITY:
Inclusion Criteria:

1. Patients >19 years old
2. Patients who underwent TAVR symptomatic severe AS
3. Provision of informed consent

Exclusion Criteria:

1. Patients requiring dual antiplatelet therapy longer than 4 weeks
2. Any conditions requiring specific antiplatelet therapy aspirin or clopidogrel
3. History of stroke or transient ischemic attack (TIA) within 6 months
4. Planned major surgery
5. Cardiogenic shock or hemodynamic instability
6. Chronic kidney disease stage 4 or 5 (eGFR <30mL/min)
7. Valve-in-valve TAVR procedure
8. Hypersensitivity or contraindication to aspirin or clopidogrel
9. Indication for anticoagulation therapy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2026-07-21 (Estimated); Study Completion 2027-07-21 (Estimated)

PRIMARY OUTCOMES:
Incidence of leaflet thrombosis | At 3 months after TAVR
  Incidence of leaflet thrombosis on cardiac CT at 3 months after TAVR

SECONDARY OUTCOMES:
Any stroke | 3 months and 6 months after TAVR
Ischemic Stroke | 3 months and 6 months after TAVR
Transient ischemic attack | 3 months and 6 months after TAVR
Thromboembolic events (composite of any stroke, myocardial infarction, systemic embolism (not involving the central nervous system), deep-vein thrombosis, or pulmonary embolism) | 3 months and 6 months after TAVR
Echocardiographic parameters (maximum and mean aortic valve pressure gradient) | at 3 months after TAVR
Echocardiographic parameters (doppler velocity index) | at 3 months after TAVR
Echocardiographic parameters (paravalvular regurgitation) | at 3 months after TAVR
Echocardiographic parameters (leaflet thrombosis) | at 3 months after TAVR
VARC-3 type 3 or 4 bleeding | 3 months and 6 months after TAVR
VARC-3 type 2 bleeding | 3 months and 6 months after TAVR

CONTACTS AND LOCATIONS:
Overall Officials: Young-Guk Ko, MD, PhD, Principal Investigator — Division of Cardiology, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No